CLINICAL TRIAL: NCT01643447
Title: A Prospective Randomized Trial Comparing Ulinastatin's Drug Protection in Hepatocellular Carcinoma(HCC)Patients'Postoperative Hepatic Failure
Brief Title: Ulinastatin Preventing Postoperative Hepatic Failure in Hepatocellular Carcinoma (HCC)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Hepatobiliary Surgery Hospital (Other)
Responsible Party: Principal Investigator, ShenFeng, director of department of special treatment, Eastern Hepatobiliary Surgery Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EHBH-RCT-2012-001
Record Dates: First submitted 2012-07-16; First posted 2012-07-18 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Ulinastatin; Hepatic Failure
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Failure | interventions — urinastatin; Glycyrrhizic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Diammonium glycyrrhizinate (Active Comparator): Conventional drugs protect liver
  Interventions: Drug: Diammonium glycyrrhizinate
- Ulinastatin (Experimental): Ulinastatin Preventing Postoperative Hepatic Failure in Hepatocellular carcinoma (HCC)
  Interventions: Drug: Ulinastatin

INTERVENTIONS:
Drug: Ulinastatin — Ulinastatin Preventing Postoperative Hepatic Failure in Hepatocellular carcinoma (HCC)
  Arms: Ulinastatin
Drug: Diammonium glycyrrhizinate
  Arms: Diammonium glycyrrhizinate

SUMMARY:
The purpose of this study is to confirm that Ulinastatin is a safe and effective drug and it can reduce the incidence of postoperative hepatic failure in HCC patients. To evaluate that Ulinastatin can improve survival in HCC patients or not.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC), a serious disease with high incidence at home and abroad, still shows a rising trend. Postoperative hepatic failure remains a major reason of liver resection's failure.

• As broad spectrum of enzyme inhibitors, Ulinastatin has the valid therapeutical effect of hepatic failure and hepatic ischemia-reperfusion injury in animal experiment. And it restrain inflammatory mediator to release. But it's lack of clinical evidence that Ulinastatin reduce the incidence of postoperative hepatic failure in HCC patients The purpose of the study is to assess the effort for comparing Ulinastatin's drug protection in patients with hepatocellular carcinoma (HCC) for postoperative hepatic failure and to evaluate that Ulinastatin can improve survival in HCC patients or not.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients > 35 years and <=55 years of age.
2. confirmed case (patients with HCC)
3. Tumors can be radical removed and resection volume was 50% to 70%.
4. Criteria of liver function: Child A level, serum bilirubin ≤ 1.5 times the upper limit of normal value,alanine aminotransferase and aspartate aminotransferase ≤ 2 times the upper limit of normal value.
5. No dysfunction in major organs; Blood routine, kidney function, cardiac function and lung function are basically normal. Hbg ≥ 90g/L, WBC ≥ 3.000 cells/mm³,platelets ≥ 80.000 cells/mm³.
6. Karnofsky Performance Score performance over 60.
7. Patients who can understand this trial and have signed information consent.

Exclusion Criteria:

1. Patients who have undergone previous treatment by Ulinastatin.
2. Patients with apparent cardiac, pulmonary, cerebronic and renal dysfunction, which may affect the treatment of liver cancer.
3. Patients with other diseases which may affect the treatment mentioned here.
4. Patients with medical history of other malignant tumors.
5. Subjects participating in other clinical trials.
6. Extrahepatic metastasis, portal vein or other major vascular involvement. liver function: Child B C.
7. Patients would not sign the consent to the trial.

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2012-05; Primary Completion 2014-12 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
the overall survival rate of each group | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Li Aijun, MD, Study Chair — Eastern Hepatobiliary Surgery Hospital, Second Military Medical University
Locations (1):
- Eastern Hepatobiliary Surgery Hospital, Shanghai, Shanghai Municipality, China